CLINICAL TRIAL: NCT03706924
Title: Open-Label, Randomized, Parallel-group, Comparative Study of Pharmacokinetics and Bioequivalence of VM-1500FDC (Viriom Ltd, Russia) and Elpida® (Viriom Ltd, Russia) and Truvada® (Gilead Sciences Ireland UC, UK) When сo-administrated Once Daily Fasting in Healthy Subjects
Brief Title: Comparative Study of PK and BE of VM-1500FDC (Fixed-dose Combination) and Elpida® With Truvada® сo-administrated 1 Daily Fasting in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HIV-VM1500FDC-01
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: HIV-1-infection
Keywords: HIV -1; elsulfavirine fixed-dose combination
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — elsulfavirine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VM-1500FDC (Experimental): VM-1500FDC (tenofovir 300 mg/elsulfavirine 20 mg/emtricitabine 200 mg), once daily fasting
  Interventions: Drug: VM-1500FDC
- Elpida® & Truvada® (Active Comparator): Elpida®, 20 mg + Truvada® (tenofovir 300 mg / emtricitabine 200 mg), once daily fasting
  Interventions: Drug: Elpida®; Drug: Truvada®

INTERVENTIONS:
Drug: VM-1500FDC — A fixed-dose combination of three active substances: tenofovir 300 mg + elsulfavirine 20 mg + emtricitabine 200 mg, film-coated tablets
  Other Names: VM1500FDC
  Arms: VM-1500FDC
Drug: Elpida® — Elpida®, capsules, elsulfavirine 20 mg
  Other Names: VM-1500; VM1500; Elsulfavirine
  Arms: Elpida® & Truvada®
Drug: Truvada® — Truvada® (tenofovir 300 mg / emtricitabine 200 mg), film-coated tablets
  Arms: Elpida® & Truvada®

SUMMARY:
Open-label, randomized, parallel-group, comparative study of pharmacokinetics and bioequivalence of VM-1500FDC (elsulfavirine/emtricitabine/tenofovir fixed-dose combination) and Elpida® with Truvada® (emtricitabine/tenofovir) co-administered by healthy male subjects. The study will also assess safety profile of study drugs.

DETAILED DESCRIPTION:
The study assesses PK and bioequivalence of the developed new drug VM-1500FDC - a fixed combination of three active substances: elsulfavirine (NNRTI), emtricitabine (NRTI) and tenofovir (NRTI) to Elpida® and Truvada® co-administered. The combination is intended for once daily administration (1 tablet) for the treatment of HIV-1 infection in adult patients. Thus, the purpose of this combination is to simplify the dosage regimen and improve patient compliance

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking male subjects between the ages of 20 and 40 years (inclusive);
2. Verified diagnosis of "healthy" according to standard clinical, laboratory and instrumental examination methods;
3. Body weight from 60 to 95 kg and Body Mass Index from 19.0 to 27.0 kg/m;
4. A negative result in tests for alcohol and drugs;
5. The subject's consent to use adequate contraception methods during the study and 3 month after end of study: condom with spermicide (foam, gel, cream, suppositories);
6. Signed the Participant Explanation Sheet and the Informed Consent Form.

Exclusion Criteria:

1. Chronic diseases of cardiovascular, bronchopulmonary, neuroendocrine, musculoskeletal system, as well as diseases of the gastrointestinal tract, liver, kidneys, blood;
2. Variables of standard laboratory and instrumental parameters are beyond the normal limits Variables of standard laboratory and instrumental parameters are beyond the normal limits (taking into account the acceptable limits of laboratory parameters);
3. Surgical interventions on the gastrointestinal tract in medical history (except appendectomy);
4. Systolic pressure less than 90 mm Mercury or above 130 mm Mercury, diastolic pressure less than 60 mm Mercury or above 85 mm Mercury, heart rate less than 60 BPM or more than 90 BPM at screening;
5. Regular intake of drugs less than 2 weeks prior to screening (including herbal preparations and dietary supplements); intake of drugs that have a pronounced effect on hemodynamics, liver function, etc. (for example, barbiturates, omeprazole, cimetidine, etc.) less than 30 days prior to screening;
6. Presence of antibodies to HIV and hepatitis C virus, presence of hepatitis В surface antigen, a positive syphilis test;
7. An unstable sleep structure (e.g., night work, sleep disorders, insomnia, recent return from another time zone, etc.), extreme physical activity (e.g. weight lifting), a special diet (e.g. vegetarian, vegan);
8. Signs of alcohol (taking more than 10 units of alcohol per week ) or drug addiction; alcohol or drugs consumption within 4 days prior to screening; cigarettes smoking 3 months prior to screening; positive drug and/or alcohol test;
9. Burdened allergic medical history (including drug intolerance and food allergy);
10. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
11. Hypersensitivity to tenofovir, elsulfavirine or emtricitabine, as well as any other component of the study drugs;
12. Blood/plasma donation (450 ml of blood or plasma and more) less than 2 months prior to screening;
13. Treatment with a study drug in framework of other clinical trials within 30 days prior to screening (including follow-up visits);
14. Acute infectious diseases less than 4 weeks prior to screening;
15. Incapable of reading or writing; no desire to understand and adhere to the study protocol procedures; non-compliance with the drugs intake regimen or execution of procedures, which as the Investigator may think may affect the study results or subject's safety and prevent the subject from further participation in the study; any other associated medical or serious psychological conditions making the subject not eligible to participate in the clinical study, restricting legality of obtaining the informed consent or affecting the subject's ability to take part in the study.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of VM1500A | 29 days
Plasma concentration of elsulfavirine | 29 days
Plasma concentration of emtricitabine | 29 days
Plasma concentration of tenofovir | 29 days

SECONDARY OUTCOMES:
Frequency and severity of AEs and SAEs | 29 days
  Frequency and severity of AE, recorded after administration of the drug according to subjective complaints, changes in vital signs, ECG, laboratory results and physical examination compared to the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Elena Mazygula, PhD, Principal Investigator — Private non - governmental health care institution "Scientific Clinical Center of the open joint - stock company Russian Railways"
Locations (2):
- Russia (2):
  - Central City Clinical Hospital Reutov, Reutov, Moscow Oblast
  - Private non - governmental health care institution "Scientific Clinical Center of the open joint - stock company Russian Railways", Moscow

IPD SHARING:
Plan to Share IPD: No